CLINICAL TRIAL: NCT05928481
Title: The Effect of Simulation-based Postpartum Hemorrhage Management on the Practice Skills, Satisfaction and Self-efficacy Levels of Midwifery Students
Brief Title: The Effect Of Sımulatıon-Based Postpartum Bleedıng Management On Mıdwıfery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SBÜ-AYDINKARTAL-001
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Postpartum Hemorrhage
Keywords: Simulation; Midwifery; Postpartum hemorrhage; Satisfaction; Self-efficacy
MeSH Terms: conditions — Postpartum Hemorrhage; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (n:39) (Experimental): Postpartum hemorrhage management practices were applied to the students in the intervention group on a high-reality Gaumard Scientific brand, product code: S550.100 Noella simulator in the simulation laboratory of the Midwifery department.
  Interventions: Other: Simulation-based postpartum bleeding management training
- Control group (n:39) (No Intervention): Postpartum hemorrhage management practices were applied to the students in the control group on a standard adult patient model in the basic skills laboratory.

INTERVENTIONS:
Other: Simulation-based postpartum bleeding management training — Postpartum hemorrhage management practices were applied to the students in the intervention group on a high-reality Gaumard Scientific brand, product code: S550.100 Noella simulator in the simulation laboratory of the Midwifery department.
  Arms: İntervention group (n:39)

SUMMARY:
This study was planned to determine the effect of simulation-based postpartum hemorrhage management on the application skills, satisfaction, self-confidence and self-efficacy-competences of Health Sciences University Hamidiye Health Sciences Faculty Midwifery Department 3rd year students. The research, which was planned in a randomized controlled experimental design, will be conducted with Istanbul Health Sciences University Hamidiye Health Sciences Faculty 3rd year midwifery (N:82) students. Students participating in the study will be divided into intervention (n:41) and control (n:41) groups according to the computer-assisted simple random sampling technique. Before the application, both groups will be given 2 hours of theoretical information on the evaluation and management of postpartum hemorrhage. 41 students assigned to the intervention group will be given a high-fidelity simulator, and 41 students assigned to the control group will be given practical training accompanied by an adult standard patient care model. "Descriptive Information Form", "Evaluation of Simulation-Based Learning Scale", "Student Satisfaction and Self-Confidence in Learning Scale", "Self-Efficacy Scale" and "Early Postpartum Hemorrhage Management Skill Evaluation Form" will be applied to the students participating in the research.

DETAILED DESCRIPTION:
This study was planned to determine the effect of simulation-based postpartum hemorrhage management on the application skills, satisfaction, self-confidence and self-efficacy-competences of Health Sciences University Hamidiye Health Sciences Faculty Midwifery Department 3rd year students.

The research population consisted of 3rd grade students who took the "Risky Birth and Postpartum Period" course, studying at the Department of Midwifery, Hamidiye Faculty of Health Sciences, in the spring semester of the 2021-2022 academic year (N:82). Students who volunteered to participate in the study were included in the study. In the study, the entire target population was reached, except for the 4 students who were absent from the "Risky Birth and Postpartum Period" course (N:78). Computer-assisted randomization will be used in the study, and random assignment was made to the intervention (n:39) and control (n:39) groups by entering the number of cases through the program whose URL address is https://www.randomizer.org.

An introductory information form was applied to all groups, and informed consent was obtained from the students before the applications. The students were given information about the introduction of the simulator and the model, the flow chart of the training plan, the content of the training plan, the environment, the locations of the materials. Before the application, all groups were given theoretical information about postpartum hemorrhage management for 2 hours with a power point presentation. "Student Satisfaction and Self-Confidence Scale in Learning" and "Self-Efficacy Scale" were applied as a pre-test after the information. Intervention group students were given practical training on postpartum hemorrhage assessment and management in the basic skills laboratory, accompanied by an adult standard patient care model, with a high-reality Gaumard Scientific brand, product code: S550.100 Noella simulator in the simulation laboratory of the Midwifery department. After the application, "Student Satisfaction and Self-Confidence in Learning Scale", "Self-Efficacy Scale" and "Early Postpartum Hemorrhage Management Skill Assessment Form" were applied to all students as a post-test, and "Scale for Evaluation of Simulation-Based Learning" to the intervention group. Four weeks after the training, the "Early Postpartum Hemorrhage Management Skill Assessment Form" and "Self-Efficacy Scale" were applied to the students again as a follow-up test.

After the research was completed, postpartum hemorrhage management was applied to the control group students with a high-reality simulator, accompanied by a scenario, so that all students could benefit from the benefits of simulation-based education. At the end of the simulation applications, an analysis session was held for the students accompanied by the video recordings taken during the applications. During the debriefing session, it was aimed to help students see their mistakes and organize their practices without judging by using a constructive language.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research.
* Being a third year student at SBU, Hamidiye Faculty of Health Sciences, Midwifery Department.
* To have successfully completed the theory and practice of basic principles and practices in midwifery.
* To have taken the risky birth and postpartum period lesson.

Exclusion Criteria:

* Not volunteering to participate in the research.
* Not to be a third year student at the Faculty of Health Sciences, Hamidiye, Department of Midwifery.
* Not having successfully completed the theory and practice of basic principles and practices in midwifery.
* Not having taken the risky birth and postpartum lesson.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 5 minutes
  In this form, which was created by the researchers based on the literature, the participants' age, the high school they graduated from, the education level of their parents, their willingness to choose the profession, their feeling of belonging to the profession, etc. questions are included.
Student Satisfaction and Self-Confidence Scale in Learning | 10 minutes
  According to the Turkish version of the scale, the total number of items is 12. This scale measures student satisfaction and self-confidence towards learning in a simulation environment. The scale consists of two sub-titles: "Satisfaction with Current Learning" and "Self-Confidence in Learning". There is no negative item in the scale. A 5-point likert expressing student feelings was used; 1) Strongly disagree, 2) Disagree, 3) Undecided, 4) Agree, and 5) Strongly Agree. Cronbach's alpha value was 0.85 for "Satisfaction with Current Learning" and 0.77 for "Self-Confidence in Learning". In the scoring of the scale, the formula of dividing the total score obtained by the answers by the number of item 33 is used. In the scoring, 1 point was determined as the lowest and 5 points as the highest. As the total score obtained from the scale increases, student satisfaction and self-confidence in learning increase.
Self-Efficacy Scale | 10 minutes
  The scale, which does not belong to any subjective domain, measures the perception of general self-efficacy and efficacy. The Self-Efficacy Scale is structured as a 5-point Likert-type scale consisting of 23 items, and a minimum of 23 and a maximum of 115 points can be obtained from the scale. For each item on the scale, one of the options 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well, is based on the score given for each item. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 on the scale are scored in the opposite direction. An increase in the total score that can be obtained from the scale indicates that the general self-efficacy-efficacy perception is high.

SECONDARY OUTCOMES:
Evaluation Scale of Simulation-Based Learning | 10 minutes
  There are 37 items in the scale, which consists of five sub-dimensions. The answers are scored in a five-point Likert type, ranging from 1 (strongly disagree) to 5 (strongly agree), and the total score varies between 37-185. All statements in the scale are positive and there is no reverse coded item. The content validity index of the scale was 0.89, the total Cronbach's alpha value was 0.95 and the Cronbach's alpha values of the sub-dimensions ranged between 0.77-0.90.
Self-Efficacy Scale | 10 minutes
  The scale, which does not belong to any subjective domain, measures the perception of general self-efficacy and efficacy. The Self-Efficacy Scale is structured as a 5-point Likert-type scale consisting of 23 items, and a minimum of 23 and a maximum of 115 points can be obtained from the scale. For each item on the scale, one of the options 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well, is based on the score given for each item. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 on the scale are scored in the opposite direction. An increase in the total score that can be obtained from the scale indicates that the general self-efficacy-efficacy perception is high.
Student Satisfaction and Self-Confidence Scale in Learning | 10 minutes
  According to the Turkish version of the scale, the total number of items is 12. This scale measures student satisfaction and self-confidence towards learning in a simulation environment. The scale consists of two sub-titles: "Satisfaction with Current Learning" and "Self-Confidence in Learning". There is no negative item in the scale. A 5-point likert expressing student feelings was used; 1) Strongly disagree, 2) Disagree, 3) Undecided, 4) Agree, and 5) Strongly Agree. Cronbach's alpha value was 0.85 for "Satisfaction with Current Learning" and 0.77 for "Self-Confidence in Learning". In the scoring of the scale, the formula of dividing the total score obtained by the answers by the number of item 33 is used. In the scoring, 1 point was determined as the lowest and 5 points as the highest. As the total score obtained from the scale increases, student satisfaction and self-confidence in learning increase.
Early Postpartum Bleeding Skill Assessment Form | 20 minutes
  The form developed by the researchers based on the literature was given its final shape in line with the opinions of twelve experts. Form; It consists of two parts, "Part I: Early Postpartum Hemorrhage Evaluation Procedure Steps" and "Part II: Behaviors to Observe in Cases of Postpartum Hemorrhage". first chapter, 30; The second part contains 25 questions and there are 55 questions in total in the scale. Scale scoring; It was made in line with the parameters "Needs to be Improved (0 Points)", "Adequate (1 Point)", "Mastered (2 points)". Bleeding management skill levels of students in the early postpartum period, skill evaluation form; the first part is a minimum of 0 points, a maximum of 60 points; the second part is a minimum of 0 points, a maximum of 50 points; their total scores were evaluated with the sum of the points they received, with a minimum of 0 points and a maximum of 110 points.

OTHER OUTCOMES:
Early Postpartum Bleeding Skill Assessment Form | 20 minutes
  The form developed by the researchers based on the literature was given its final shape in line with the opinions of twelve experts. Form; It consists of two parts, "Part I: Early Postpartum Hemorrhage Evaluation Procedure Steps" and "Part II: Behaviors to Observe in Cases of Postpartum Hemorrhage". first chapter, 30; The second part contains 25 questions and there are 55 questions in total in the scale. Scale scoring; It was made in line with the parameters "Needs to be Improved (0 Points)", "Adequate (1 Point)", "Mastered (2 points)". Bleeding management skill levels of students in the early postpartum period, skill evaluation form; the first part is a minimum of 0 points, a maximum of 60 points; the second part is a minimum of 0 points, a maximum of 50 points; their total scores were evaluated with the sum of the points they received, with a minimum of 0 points and a maximum of 110 points.
Self-Efficacy Scale | 10 minutes
  The scale, which does not belong to any subjective domain, measures the perception of general self-efficacy and efficacy. The Self-Efficacy Scale is structured as a 5-point Likert-type scale consisting of 23 items, and a minimum of 23 and a maximum of 115 points can be obtained from the scale. For each item on the scale, one of the options 1-Does not describe me at all, 2-Describes me a little, 3-I am undecided, 4-Describes me well, 5-Describes me very well, is based on the score given for each item. Items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16, 17, 18, 20, and 22 on the scale are scored in the opposite direction. An increase in the total score that can be obtained from the scale indicates that the general self-efficacy-efficacy perception is high.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No